CLINICAL TRIAL: NCT03898505
Title: Clinical Investigation on the Safety of Avocado Pulp Lipids
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Guelph (Other)
Collaborators: Advanced Orthomolecular Research (Unknown)
Responsible Party: Principal Investigator, Paul A. Spagnuolo, Associate Professor, University of Guelph
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 232024
Record Dates: First submitted 2019-03-29; First posted 2019-04-02 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Obesity; Avocado; Overnutrition; Nutritional Disorder; Metabolic Disease; Lipid Metabolism Disorders
Keywords: Avocado; Polyhydroxylated Fatty Alcohols; Avocatin B
MeSH Terms: conditions — Obesity; Overnutrition; Nutrition Disorders; Metabolic Diseases; Lipid Metabolism Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo powder containing only non-medicinal ingredients used in the test product: Oryza sativa (rice) bran extract (65-70% w/w of total placebo formulation), sodium bicarbonate, rosemary extract, xylitol, silicon dioxide, microcrystalline cellulose, rice hull powder, strawberry flavour. Participants in the placebo group will ingest 1 scoop of the placebo material per day (30-35g). Placebo powder is to be dissolved/blended in 12-16 ounces of a smoothie like diluent (e.g., 2% milk (with or without lactose), soy milk, coconut milk, or fruit juice of the participant's choice) and consumed orally. Placebo will be consumed once per day for 60 days.
  Interventions: Other: Placebo
- Low Dose (Experimental): All Participants randomized to the low dose group will be consuming food grade avocado pulp powder (AvoMax) that will deliver a 50 mg dose of bioactive polyhydroxylated fatty alcohols (PFAs), avocadyne and avocadene. Participants in the low dose group will ingest 1 scoop of this test product per day (30-35g). Low dose test product is to be dissolved/blended in 12-16 ounces of a smoothie like diluent (e.g., 2% milk (with or without lactose), soy milk, coconut milk, or fruit juice of the participant's choice) and consumed orally. Low dose test product will be consumed once per day for 60 days.
  Interventions: Dietary Supplement: AvoMax (Low Dose)
- High Dose (Experimental): All Participants randomized to the high dose group will be consuming food grade avocado pulp powder (AvoMax) that will deliver a 200 mg dose of bioactive polyhydroxylated fatty alcohols (PFAs), avocadyne and avocadene. Participants in the high dose group will ingest 1 scoop of this test product per day (30-35g). High dose test product is to be dissolved/blended in 12-16 ounces of a smoothie like diluent (e.g., 2% milk (with or without lactose), soy milk, coconut milk, or fruit juice of the participant's choice) and consumed orally. High dose test product will be consumed once per day for 60 days.
  Interventions: Dietary Supplement: AvoMax (High Dose)

INTERVENTIONS:
Dietary Supplement: AvoMax (Low Dose) — AvoMax (Low Dose) is a natural spray-dried avocado powder, which contains 50 mg of a combination of bioactive polyhydroxylated fatty alcohols (PFAs), avocadyne and avocadene.
  Arms: Low Dose
Dietary Supplement: AvoMax (High Dose) — AvoMax (High Dose) is a natural spray-dried avocado powder, which contains a total of 200 mg of a combination of bioactive polyhydroxylated fatty alcohols (PFAs), avocadyne and avocadene.
  Arms: High Dose
Other: Placebo — Placebo product is powder containing only non-medicinal ingredients used in the test product: Oryza sativa (rice) bran extract (65-70% w/w of total placebo formulation), sodium bicarbonate, rosemary extract, xylitol, silicon dioxide, microcrystalline cellulose, rice hull powder, strawberry flavour.
  Arms: Placebo

SUMMARY:
Obesity and diabetes are a significant global burden and there is an immediate need for novel treatments and management strategies. Our laboratory determined that avocado derived 17 carbon polyhydroxylated fatty alcohols (PFAs) are inhibitors of fatty acid oxidation (FAO) that impart minimal toxicity in mice. FAO is altered in numerous disease states including obesity and diabetes. In these chronic diseases, excessive FAO in muscle and liver mitochondria cause metabolic overload and inefficiency which drives obesity-associated glucose intolerance and insulin insensitivity. The increased FAO that occurs in obese and diabetic individuals depletes several substrates and intermediates of the Krebs cycle, making them less efficient at using oxidative phosphorylation for energy, which can ultimately lead to glucose insensitivity and weight gain. For these reasons, inhibition of FAO is now an established therapeutic approach for the treatment of type II diabetes as reducing FAO: i) improves cellular metabolism to shift towards the more thermogenic oxidative phosphorylation and glycolysis, and ii) reduces hyperglycemia via inhibiting liver gluconeogenesis while improving glucose homeostasis.

In collaboration with an industry partner, Advanced Orthomolecular Research (AOR; Calgary, AB), the investigators have developed a supplement containing a blend of 17-carbon PFAs found inside a commercially available food grade avocado powder. The primary objective of this clinical trial is to determine if the avocado derived supplement is safe for oral consumption compared to a placebo-controlled group.

DETAILED DESCRIPTION:
This is a single center, double-blind, placebo-controlled, randomized clinical trial. 30 healthy subjects are planned. After screening and recruitment, subjects will be randomly allocated to treatment groups (low dose avocado powder or high dose avocado powder) or placebo control group. Once recruitment, randomization, baseline measurements as well as treatment allocation is completed (on the first site visit), each subject will orally consume one scoop (30-35g of material) of the avocado supplement, blended in 12-16 ounces of a smoothie like diluent, once per day for 60 days. The placebo group will also consume one scoop (30-35g of material) containing only non-medicinal ingredients used in the test product. Primary and secondary endpoint evaluations will be taken at baseline (site visit 2), day 30 (site visit 3) and day 60 (site visit 4) at each of the 3 study site visits as well as via weekly telephone calls to participants. Total duration of subject participation will be 60 days. Total duration of the study is expected to be 61 days.

ELIGIBILITY:
Inclusion Criteria:

* adults 18 to 60 years of age
* includes non-pregnant, non-breastfeeding women on adequate birth control
* stable body weight (BMI: 18.5-29.9)
* written informed consent obtained from subject and ability for subject to comply with the requirements of the study.

Exclusion Criteria:

* Pregnant or breastfeeding
* History or presence of diabetes
* History or presence of hypertension
* History or presence of dyslipidemia
* History or presence of major depressive disorders
* History or presence of chronic liver disorders
* History or presence of kidney disorders
* History or presence of blood disorders
* Previous bariatric surgery (or any major surgeries or medical procedures to be scheduled within the time frame of the study)
* Use of medication that causes significant weight gain or loss
* Allergies to or inhibitions consuming all three choices of: 2% lactose free milk, soy milk, or coconut milk
* Allergies to any ingredients in the placebo/investigational product
* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-11-24 (Actual); Primary Completion 2018-06-25 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of Adverse Events (AE) | During treatment period (Day 1 to Day 60)
  Number of treatment emergent adverse events according to CTCAE v5.0.

SECONDARY OUTCOMES:
Hematology | At screening and during treatment period (day 30 and day 60)
  Number of clinically relevant changes in hematology markers as assessed by: hematocrit (HCT), hemoglobin (Hb), red blood cell count (RBC), mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), mean corpuscular hemoglobin concentration (MCHC), white blood cell count (WBC), differential blood count (neutrophils, lymphocytes, monocytes, eosinophils and basophils), reticulocytes absolute count, and mean platelet volume (MPV). Assessments will be performed at screening and during treatment period.
Biochemistry | At screening and during treatment period (day 30 and day 60)
  Number of clinically relevant changes in serum biochemistry. Enzymes: alanine transaminase, creatine phosphokinase. Substrates: bilirubin (total), creatinine. Assessments will be performed at screening and during treatment period.
Glycated Hemoglobin (HbA1c) | At screening and during treatment period (day 30 and day 60)
  Mean absolute glycated hemoglobin (HbA1c) change from baseline
Body Weight | At screening and during treatment period (day 30 and day 60)
  Mean absolute body weight change from baseline
Body Mass Index (BMI) | At screening and during treatment period (day 30 and day 60)
  Mean absolute body mass index (BMI) change from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Paul Spagnuolo, PhD, Principal Investigator — University of Guelph; Mary M Warndl, MD, Study Chair — Medical Monitor; Kim Bretz, ND, Study Director — Fundamentals of Health Naturopathic Medicine Clinic; Nawaz Ahmed, MSc, Study Director — University of Guelph
Locations (1):
- Fundamentals of Health Naturopathic Medicine Clinic, Waterloo, Ontario, Canada